CLINICAL TRIAL: NCT06070688
Title: Does an Adjunct Diagnostic Test That Can Discriminate Bacterial From Viral Etiology Early in the Management of Respiratory Infections Improve Management Accuracy and Quality in the Acute Care Setting?
Brief Title: An Adjunct Test Distinguishing Bacterial From Viral Etiology Improves Resource Utilization and Efficiency in the ED.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: MeMed Diagnostics Ltd. (Industry)
Responsible Party: Principal Investigator, David Robinson, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HSC-MS-23-0692
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Tract Infections
Keywords: bacterial infection; viral infection
MeSH Terms: conditions — Respiratory Tract Infections; Bacterial Infections; Virus Diseases

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Statistician assessing financial and resource utilization between study arms (primary and secondary outcomes) will be blinded as to which cohort had the results of the Memed diagnostic test (experimental vs standard groups)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MeMed BV® biomarker test and standard of care (Experimental): In addition to the standard of care for acute respiratory infections, the experimental arm shall reveal the results of the 'BV' test to the clinician co-investigators. The BV test reports a clinical score from 1-100 that as an adjunct to usual care, may help the clinician better direct appropriate resources towards the patient.
  Interventions: Diagnostic Test: MeMed BV® biomarker test; Diagnostic Test: Usual care
- Usual Care (Active Comparator): The co-investigators shall evaluate, diagnose and manage the acute respiratory infection presenting to the ED using the standard practice known in the community. This may include hospital sepsis practice protocols, clinical judgement, and national or local practice standards.
  Interventions: Diagnostic Test: Usual care

INTERVENTIONS:
Diagnostic Test: MeMed BV® biomarker test — one purple top tube of whole blood (2-3 cc) to be used for the MeMed Key® device processing without the need for centrifuge. The MeMed BV® test takes approximately 15 minutes to process and result. After, the sample has been processed and the MeMed BV® test has resulted, the sample of blood will be discarded for each patient enrolled in the study.
  Arms: MeMed BV® biomarker test and standard of care
Diagnostic Test: Usual care — Usual care includes diagnostic hematology, chemistry, biomarkers, and culture results along with imaging, consults, and medications, in the treatment of acute viral and/or bacterial illness.

SUMMARY:
The purpose of this study is to evaluate overall changes in patient management and longer-term resource utilization between control and test arms, including (but not limited to) additional work-up (including other diagnostic tests and consults), antimicrobial treatments, disposition decisions and hospital length of stay (LOS)

DETAILED DESCRIPTION:
The trial seeks to compare the benefits of adding a diagnostic test that can distinguish the etiology of an acute respiratory illness early in the work-up and management. All adult patients shall be evaluated through the Emergency Department (ED) as an undiagnosed acute reparatory illness (URI). The included patient cohort must present with SIRS criteria and be ill enough to require immediate blood draw and management by the ED. Excluded are any URIs with a predetermined diagnosis or subjects presenting with illness not determined to be a URI as a primary diagnosis. The experimental arm of the study shall have in addition to the standard of care labs and diagnostics, a novel protein array blood test that can distinguish bacterial from viral disease. The control group will not receive these results. The trial seeks to examine the difference in clinical outcomes when a adjunct biomarker than can help the clinician guide more accurate therapy is available early in the diagnostic workup. Benefits are defined in the primary and secondary outcomes as reduced resources expended through reduced laboratory, radiological, blood bank, and pharmaceutical expenditures. Comparative resource utilization costs include changes in hospital and or ED length of stay, lower follow up visits and readmissions, less inpatient and outpatient physician consultants and services called for to manage the patients care, and overall costs. Both primary and secondary outcomes will be used to categorize the costs and resources required to manage the patient. Primary objective is to evaluate overall changes in patient management and longer-term resource utilization between control and test arms, including (but not limited to) additional work-up (including other diagnostic tests and consults), antimicrobial treatments, disposition decisions and hospital length of stay (LOS). The exploratory objective is to evaluate changes between control and test arm in ED LOS, bounce backs (patients returning within 72 hours), work-up costs and the impact of physician seniority.

ELIGIBILITY:
Inclusion Criteria for main study population :

* Current disease duration ≤ 7 days
* Temperature ≥ 37.8°C (100°F) or tactile fever, noted at least once within the last 7 days
* Clinical suspicion of bacterial or viral respiratory tract infection (RTI)

Exclusion Criteria for main study population:

* Systemic antibiotics taken up to 48 hours prior to presentation
* Outpatient steroids taken within 48 hours prior to presentation
* Suspicion and/or confirmed diagnosis of infectious gastroenteritis/colitis
* Inflammatory disease
* Congenital immune deficiency (CID)
* A proven or suspected infection on the presentation with Mycobacterial, parasitic or fungal (e.g., Candida, Histoplasma, Aspergillus) pathogen
* Human immunodeficiency virus(HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (self-declared or known from medical records)
* Major trauma and/or burns in the last 7 days
* Major surgery in the last 7 days
* Pregnancy - Self reported or medically confirmed
* Active malignancy - Cancer diagnosed within the previous six months, recurrent, regionally advanced, or metastatic cancer, cancer for which treatment had been administered within six months, or hematological cancer that is not in complete remission.
* Current treatment with immune-suppressive or immune-modulating therapies, at some point in the past 10 days
* Hemodynamically unstable (require life-saving interventions such as vasopressors)
* Patients transferred from another facility who already have a differentiated respiratory illness (known diagnosis e.g., culture positive results)
* Consider unsuitable for the study by the study team

Inclusion Criteria for Subgroup:

* Written informed consent must be obtained from the patient or his/her legal guardian
* Current disease duration ≤ 7 days
* Clinical suspicion of bacterial or viral sepsis based on 2 or more SIRS criteria OR Clinical suspicion of bacterial or viral respiratory tract infection (RTI) AND temperature ≥ 37.8°C (100°F) or tactile fever, noted at least once within the last 7 days

Patients fulfilling one or more of the following exclusion criteria from the main group are eligible for the subgroup cohort:

* Systemic antibiotics taken up to 48 hours prior to presentation
* Outpatient steroids taken within 48 hours prior to presentation
* Suspicion and/or confirmed diagnosis of infectious gastroenteritis/colitis
* Inflammatory disease (e.g., IBD, SLE, RA, other vasculitis)
* Congenital immune deficiency (CID)
* A proven or suspected infection on the presentation with Mycobacterial (e.g., MAC, MABC), parasitic or fungal (e.g., Candida, Histoplasma, Aspergillus) pathogen
* HIV, HBV, or HCV infection (self-declared or known from medical records)
* Major trauma and/or burns in the last 7 days
* Major surgery in the last 7 days
* Pregnancy - Self reported or medically confirmed
* Active malignancy of a solid tumor - Cancer diagnosed within the previous six months, recurrent, regionally advanced, or metastatic cancer, cancer for which treatment had been administered within six months, or hematological cancer that is not in complete remission
* Current treatment with immune-suppressive or immune-modulating therapies, at some point in the past 10 days
* Hemodynamically unstable (require life-saving interventions such as vasopressors)
* Patients transferred from another facility who already have a differentiated respiratory illness (known diagnosis e.g., culture positive results)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cost of any additional diagnostic tests done by a participant | from day of admission to emergency department upto about 28 day follow up
  Additional diagnostic tests may include serial complete blood count (CBC)s, additional blood cultures, viral cultures and serial basic metabolic panel (BMP) blood bank
Cost of any additional consults done by a participant | from day of day of admission to emergency department upto about 28 day follow up
  Comparative metric between the experimental and control groups
Total cost of any antimicrobial treatments by a participant | end of study (about 28 days from baseline)
  Comparative metric between the experimental and control groups
Number of participants that were admitted to the hospital | end of study (about 28 days from baseline)
  Comparative metric between the experimental and control groups
Cost of hospital stay | end of study (about 28 days from baseline)
  Total costs defined as all costs including lab and diagnostic services, blood bank, pharmaceuticals, nursing, consultants, and all other services listed in the patient's work-up. Comparative metric between the experimental and control groups
Length of hospital stay | at time of discharge( from 28 days- 6months from baseline)
  Comparative metric between the experimental and control groups

SECONDARY OUTCOMES:
Length of stay in emergency department | at time of discharge from emergency department (upto about 48 hours form admission)
  Comparative metric between the experimental and control groups
Number of participants that had a bounce back as defined as patients returning any time during the 28-day call back period | end of study (about 28 days from baseline)
  Bounce backs are defined as any return to a health care entity during the 28 day period after discharge from the index visit. Comparative metric between the experimental and control groups
Emergency room work-up costs | at time of discharge from emergency department (upto about 48 hours form admission)
  Comparative metric between the experimental and control groups
Number of participants with medical interventions such as blood draws, consults and imaging used during the patient's time in the study | end of study (about 28 days from baseline)
  Comparative metric between the experimental and control groups
Quality of care as determined by the number of acute respiratory ill patients with bacterial etiology that received appropriate antibiotics | Within 1-3 hours of admission to emergency department
  Comparative metric between the experimental and control groups
Number of participants within the upper respiratory infection (URI) cohort without a bacterial source (viral, inflammatory, etc.) who appropriately did not receive antibiotics or whose antibiotic course was withheld during the patient's time in the study | end of study (about 28 days from baseline)
  Comparative metric between the experimental and control groups

CONTACTS AND LOCATIONS:
Overall Officials: David Robinson, MD,MS,MMM, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No